CLINICAL TRIAL: NCT00048334
Title: Phase I Trial of Romidepsin Given on Days One, Three, and Five in Patients With Thyroid and Other Advanced Cancers
Brief Title: Depsipeptide to Treat Thyroid and Other Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030030; 03-C-0030; NCT00052767 (obsolete NCT alias)
Record Dates: First submitted 2002-10-29; First posted 2002-10-30 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-01-07

CONDITIONS: Neoplasms
Keywords: Histone Acetylation; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Depsipeptides; romidepsin

INTERVENTIONS:
Drug: Depsipeptide, FR901228, FK228

SUMMARY:
This phase I study will evaluate the experimental drug Romidepsinin patients with advanced cancer. The study will: 1) determine how well patients tolerate Romidepsin; 2) measure blood levels of Romidepsin during treatment; 3) analyze the cellular and molecular effects of the drug; and 4) determine if Romidepsin can shrink tumors. Romidepsin has been shown to kill cancer cells growing in the laboratory and to shrink tumors in animals with various tumor types. In preliminary studies, several patients with a type of lymphoma and one patient with kidney cancer responded to treatment.

Patients 18 years of age and older with advanced cancer (excluding acute leukemia) may be eligible for this study. Candidates are screened with a medical history and physical examination, x-rays and CT scans, and blood and urine tests. Patients with thyroid cancer may also have magnetic resonance imaging (MRI). This test uses a magnetic field instead of x-rays to obtain images or body organs and tissues.

Participants receive three infusions of Romidepsin administered through an intravenous line over 4 hours on days 1, 3 and 5 of a 21-day treatment cycle. The intravenous line is a catheter (plastic tube) placed in a vein and may be a peripheral line, inserted in a vein in the arm, or a central line, in which the tube is placed under the skin of the chest or neck into a major vein. Patients are hospitalized for the first 6 days of the first cycle to monitor heart rate. Those who tolerate the treatment well may continue as an outpatient.

In addition to drug therapy, participants undergo the following procedures:

* Blood tests: Small amounts of blood are drawn frequently during the first five days of treatment to measure Romidepsin levels and to see how the body uses and excretes the drug. A heparin lock (an indwelling device to keep the vein open) may be put in the vein to prevent the need for repeated needle sticks.
* Biopsies (removal of a small sample of tumor tissue): Tumors that are accessible may be biopsied at the start of the study and at different times during treatment. Biopsies are done no more than three times per cycle, and no more than nine biopsies are done within a year. The samples are examined for the effects of Romidepsin on proteins that control the way cells divide and stay alive.
* Apheresis: This procedure is done to collect white blood cells and cancer cells for research. Blood is collected through a needle in an arm vein and directed into a machine that separates it into its components by centrifugation (spinning). The white cells are removed and the red cells are returned to the patient through the same needle or through another needle in the other arm.
* Scans and x-rays: Imaging studies are usually done before starting treatment. Some of them are repeated at every 2 cycles (6 weeks), and some at the end of the patient's participation in the study. The tests may include chest x-rays, plain x-rays of affected bones, CT scans of the chest, abdomen, and pelvis, bone scans, and a MUGA scan (special X-ray of the heart) or echocardiogram (ultrasound of the heart) to test heart function before and during the study. MRI or positron emission tomography (PET) scans may also be done to detect tumors. PET scans use a small amount of a radioactive substance injected into a vein. The radioactivity is detected by a special camera during scanning to detect cancer cells.
* Other tests include an electrocardiogram (recording of the electrical activity of the heart) before and after each dose of depsipeptide. Eye exams are done if there are vision changes or if the doctor recommends an eye test.

DETAILED DESCRIPTION:
BACKGROUND:

Romidepsin (NSC 630176, FR901228, FK228, formerly referred to as depsipeptide) is a histone deacetylase inhibitor with potent cytotoxic activity against human tumor cell lines and in vivo efficacy against both human tumor xenografts and murine tumors (1-3).

Laboratory studies suggest that longer exposure to non-toxic doses of romidepsin can enhance its molecular effects to a greater degree than short toxic doses that rapidly cause cell death.

NIS is responsible for enabling uptake of RAI in thyroid cancer, with decreased levels in tumors resistant or refractory to RAI therapy.

Our group has demonstrated that NIS expression is upregulated by romidepsin, resulting in increased sensitivity to RAI.

OBJECTIVES:

To determine the MTD of romidepsin when administered on days 1, 3 and 5.

To examine the effect of a multi-day regimen of romidepsin on surrogate markers and the expression of molecular targets.

To determine whether thyroid cancers that do not have detectable uptake of RAI will have detectable uptake after treatment.

ELIGIBILITY:

* Age 18 and over
* Evaluable disease
* Performance status ECOG 0-2
* Excluding patients that are pregnant, HIV positive, have CNS metastasis, or acute leukemia
* Left ventricular ejection fraction within normal limits. Additional cardiac criteria are noted in protocol

DESIGN:

* Phase I
* Romidepsin administered as a 4-hour intravenous infusion on days 1, 3 and 5
* Dose escalation
* Enrollment of additional cohort of 10 patients with thyroid cancer at MTD

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have histologic or cytologic confirmation of cancer (excluding acute leukemia) for which there is no known standard therapy capable of extending life expectancy.
  2. Patients must:
* Be age greater than or equal to 18 years.
* Have evaluable disease.
* Have a performance status of ECOG 0-2.
* Have no serious or intercurrent illness that can not be medically controlled and have a have a life expectancy of greater than 12 weeks.
* Give written informed consent.
* Be willing to return to National Cancer Institute for follow-up.
* Female patients of childbearing potential must have a negative pregnancy test within 1 week and must use effective contraception (hormonal or barrier methods) while being treated on protocol.

  3. Laboratory values:
* Within 7 days prior to registration: absolute neutrophil count greater than or equal to 1000/microL, platelets greater than or equal to l00,000/microL, bilirubin (total and direct) less than or equal to 1.5x upper limit of normal, and AST less than or equal to 3x upper limit of normal, creatinine less than or equal to1.5x upper limit of normal, or documented creatinine clearance of greater than or equal to 60mL/min.
* Within 4 weeks of registration: ejection fraction of greater than 50% by echocardiogram or cardiac MRI, or 45% by MUGA scan.

  4. Criteria for cohort of patients with RAI refractory non-medullary thyroid cancer to be enrolled after the MTD has been defined:
* Non-medullary thyroid carcinoma.
* progressive disease following total or near-total thyroidectomy and RAI therapy.
* Documented evidence of no, or minimally ( faint ), RAI uptake on RAI whole body scan.
* no RAI therapy within 3 months prior to study entry.
* no history of administration of IV iodinated contrast or other large iodine loads (i.e. CT, amiodarone, SSKI) during the previous 3 months.
* 24 hr urinary iodine values less than or equal to150 microg/day.

EXCLUSION CRITERIA

1. Patients with unconfirmed diagnosis will be excluded.
2. Prior or concurrent malignancies that have not been curatively treated.
3. Current or previous CNS metastasis.
4. Chemotherapy within 4 weeks, 6 weeks for nitrosoureas or mitomycin C, and 8 weeks for UCN-01.
5. HIV seropositivity.
6. Pregnant or breast-feeding patients.
7. Uncontrolled infection.
8. Patients with the following cardiac risk factors will be excluded from the study:

   * Patients with known cardiac abnormalities such as: Congenital long QT syndrome and -QTc interval greater than 480 milliseconds
   * Patients who have had a myocardial infarction within 12 months of study entry.
   * Patients who have active coronary artery disease, e.g. angina as defined by Canadian Class II-IV
   * Patients with an ECG recorded at screening showing evidence of cardiac ischemia (ST depression of greater than or equal to 2 mm).
   * Any patient in whom coronary artery disease is suspected should be referred for a cardiology consultation and if active myocardial ischemia is demonstrated, the patient should be excluded. If a noninvasive imaging study is equivocal, it may be necessary to proceed to coronary angiography.
   * Patients with congestive heart failure that meets NYHA Class II to IV definitions and/or ejection fraction less than 45% by MUGA scan or less than 50% by echocardiogram and/or MRI.
   * Patients with a history of sustained VT, VF, Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD). Patients with a history of arrhythmia should have Holter monitoring and evaluation by cardiology.
   * Patients with dilated, hypertrophic, or restrictive cardiomyopathy from prior treatment or other causes (in doubt, see ejection fraction criteria above). Patients with left ventricular hypertrophy should be discussed with the Principal Investigator or Study Chairman.
   * Patients with uncontrolled hypertension, i.e. SBP greater than or equal to 160 mm Hg or DBP greater than or equal to 95 mm Hg.
   * Patients with cardiac arrhythmia requiring anti-arrhythmic medication other than beta blocker or calcium channel blocker. Patients in whom digitalis cannot be discontinued are excluded from study.
   * Patients with Mobitz II second degree heart block who do not have a pacemaker. Patients with first degree or Mobitz I second degree heart block, bradyarrhythmias or sick sinus syndrome require Holter monitoring and evaluation by cardiology.
   * Patients with other cardiac disease may be excluded at the discretion of the PI following consultation with cardiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-10-26; Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-01 (Actual)

PRIMARY OUTCOMES:
To define the MTD of romidepsin when administered on a multi-daly regimen of days 1, 3, and 5.

SECONDARY OUTCOMES:
To correlate laboratory assays of the molecular effects of romidepsin with the administered dose.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Piekarz, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ueda H, Nakajima H, Hori Y, Fujita T, Nishimura M, Goto T, Okuhara M. FR901228, a novel antitumor bicyclic depsipeptide produced by Chromobacterium violaceum No. 968. I. Taxonomy, fermentation, isolation, physico-chemical and biological properties, and antitumor activity. J Antibiot (Tokyo). 1994 Mar;47(3):301-10. doi: 10.7164/antibiotics.47.301. PMID 7513682
- [Background] Ueda H, Manda T, Matsumoto S, Mukumoto S, Nishigaki F, Kawamura I, Shimomura K. FR901228, a novel antitumor bicyclic depsipeptide produced by Chromobacterium violaceum No. 968. III. Antitumor activities on experimental tumors in mice. J Antibiot (Tokyo). 1994 Mar;47(3):315-23. doi: 10.7164/antibiotics.47.315. PMID 8175484
- [Background] Ueda H, Nakajima H, Hori Y, Goto T, Okuhara M. Action of FR901228, a novel antitumor bicyclic depsipeptide produced by Chromobacterium violaceum no. 968, on Ha-ras transformed NIH3T3 cells. Biosci Biotechnol Biochem. 1994 Sep;58(9):1579-83. doi: 10.1271/bbb.58.1579. PMID 7765477